CLINICAL TRIAL: NCT02574247
Title: Role of the Auditory Efferent System in Auditory Perceptual Learning
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI change of institution
Sponsor: VA Loma Linda Health Care System (U.S. Federal Agency)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Ian B. Mertes, PhD, AuD, Principal Investigator, VA Loma Linda Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1137; 1F32DC015149-01 (NIH)
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Auditory Training and Auditory Efferent System
Keywords: Audiology; Auditory Pathways; Auditory Perception; Brain Stem; Cochlea; Ear, Inner; Efferent Pathways; Hair Cells, Auditory, Outer; Learning; Neurons, Efferent; Speech Perception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Training (Experimental): Participants in the Training arm will undergo 15 hours of computerized auditory training across 10 laboratory visits. Medial olivocochlear reflex function and speech perception abilities will be measured before, during, and after the training visits to examine the changes in the measurements across time.
  Interventions: Procedure: Computerized auditory training
- Control (No Intervention): Participants in the Control arm will undergo the same number of visits as the Training arm, but will not participate in computerized auditory training. Medial olivocochlear reflex function and speech perception abilities will be measured at each visit to establish the test-retest reliability of these measurements in the absence of any training.
- Speech Group (No Intervention): Participants in the Speech Group will undergo 1 visit. Medial olivocochlear reflex function and speech perception abilities will be measured at this visit to establish the correlation between these measures in the absence of any training.

INTERVENTIONS:
Procedure: Computerized auditory training — 10 sessions of computerized auditory training (1.5 hr/session) across a 15-week span.
  Arms: Training

SUMMARY:
The purpose of this study is to determine how changes in speech perception resulting from a computerized auditory training program are related to concurrent changes in auditory brainstem function resulting from the training. It is hypothesized that the degree of improvement in speech perception will be correlated with the degree of change in brainstem function.

DETAILED DESCRIPTION:
The goal of this study is to determine the impact of an auditory training program on the function of the inner ear and auditory brainstem. In normal-hearing individuals, the medial olivocochlear (MOC) branch of the auditory efferent system appears to aid with hearing signals in noise. A previous study in young normal-hearing adults found that auditory training strengthened the function of the MOC system in some participants in a way that coincided with their improvements in perceiving speech sounds in background noise. The MOC function measured at baseline also predicted the amount of success from the auditory training. Although these results are promising, it is not known if they generalize to populations that often have hearing-in-noise problems such as older and hearing-impaired adults.

This study will examine how an auditory training program impacts MOC activity in a group of older adults with normal hearing or mild hearing loss. This is a prospective study utilizing a repeated-measures design. Participants will participate in a computerized auditory training program taking place over 15 weeks. Transient-evoked otoacoustic emissions (TEOAEs) will be used to measure the strength of MOC activity at each visit. Performance on untrained stimuli (words and sentences) will also be measured. A control group (no auditory training) will also be used to establish test-retest reliability for TEOAE measurements and performance on the word and sentence testing. The results of this study may contribute to the improved diagnosis and treatment of hearing-in-noise problems in Veterans and in the civilian population.

This is a single-site study that will take place at the Auditory Research Laboratory, located at the VA Loma Linda Healthcare System (VALLHS) in Loma Linda, California. Veterans and non-Veterans, both males and females, between the ages of 35 and 89 with either normal hearing or mild sensorineural hearing loss will participate. Women and minorities will be encouraged to participate. Up to 200 volunteers will be enrolled in the study. Each eligible participant will participate in a maximum of 14 study visits.

Participants will be randomly assigned a priori to either the experimental group (auditory training) or Control group (no auditory training) using simple random assignment. Because this study will detect whether or not significant changes in MOC activity and speech perception across time occurred as a result of auditory training, the Control group is needed to establish the test-retest reliability of our outcome measures in the absence of any training.

Preliminary analyses of the data showed an association between a measure of speech perception and the strength of the efferent system. To increase statistical power in examination of this association, an additional group (Speech Group) is incorporated that includes subjects that only participate in one session, with only the measurements of speech recognition and medial olivocochlear reflex activity. The Speech Group will be assigned by the investigators.

This study consists of one experiment that will last 3 years total. Each participant in the Experimental and Control groups will participate in 12 study visits, ideally over a 15-week period. However, we will allow for the visits to take place across a 1-year period to account for participants needing to miss or reschedule some visits. We will also allow 2 additional make-up visits for each participant (for a total of 14 visits), should they need to end an experimental session early. All study visits will last between 2-3 hours. Thus, the maximum amount of participation for each participant is 52 hours (14 visits x 3 hours per visit) across a 1-year period.

Standard-of-care screenings and experimental testing will be carried out in a double-walled sound-isolated audiometric chamber adjoined to a single-walled room in the Auditory Research Laboratory, located at the VALLHS. Initial audiometric testing using standard-of-care procedures will be conducted to verify eligibility for the study and will be carried out using standard clinical equipment.

Experimental tests will consist of Transient Evoked Otoacoustic Emissions (TEOAE) testing, word/sentence recognition testing, and an auditory training program (only participants in the Experimental group will undergo the auditory training). For TEOAE testing, the basic task of the participants is similar to TEOAE procedures used clinically to evaluate hearing function objectively. Testing involves listening to sounds presented through earphones while seated comfortably in a sound-treated booth, and remaining alert but quiet in order to successfully measure responses from the cochlea and brainstem. All stimuli will be presented at moderate volumes that are well below sound levels considered hazardous by Occupational Safety and Health Adminstration (OSHA) and NIOSH standards. TEOAE measurements consist of waveforms, which are changes in sound amplitude across time.

Word/sentence testing involves listening to words and sentences presented through earphones while seated in the sound-treated booth. Speech stimuli will be presented in the presence of background noise. Participants make a response about the word(s) they heard. Sounds will be presented at safe and comfortable levels.

For the auditory training program, listeners will be seated comfortably in the sound booth at a workstation with a computer screen, keyboard, and mouse. Sounds will be presented to the participants through insert earphones. Participants will make their responses concerning what they heard by mouse click or keyboard entry. The auditory training program consists of a curriculum of word and sentence presentations in various noise levels, and performance on repeated measurements are tracked throughout the subject's participation in the program.

This is a minimal risk study. The participants will all be healthy adults (other than mild hearing loss in some participants). There are no foreseeable risks involved in these studies beyond those associated with routine audiological practice, such as boredom or fatigue during testing. All sound levels to be used in the study fall below the Damage Risk Criteria established by OSHA for intensity-duration interaction.

Participants will be provided with as many breaks during testing as they or the experimenter feel are helpful to minimize mental fatigue and boredom. Loudness levels of stimuli are carefully controlled, with frequent calibration and monitoring of laboratory equipment. Participant confidentially will be protected by using only participant codes (three numbers) to label data collection sheets and computer data files. All data records will be stored on password-protected computers or as hard copy in locked offices or laboratories. Participant safety and comfort and data collection will be constantly monitored for each participant by the research team member collecting the data for that participant. Overall data collection will be monitored by the Principal Investigator. Following completion of the study, all data will be maintained in accordance with Veterans Health Administration guidelines.

Regarding potential benefits of participating, all participants will receive an up-to-date hearing screening and a further understanding of their own hearing. Participants in the Experimental group may or may not notice an improved ability to hear sounds in background noise after undergoing auditory training. The knowledge gained from this study may also benefit individuals with hearing-in-noise problems by contributing to improved diagnosis and treatment of hearing-in-noise problems in Veterans and in the civilian population.

ELIGIBILITY:
Inclusion Criteria:

* 3-frequency pure-tone average ≤40 decibels hearing level (dB HL)
* Air-bone gaps ≤10 decibels (dB) from 500-4000 Hz
* 226-Hz tympanograms within normal limits
* Measurable acoustic reflexes bilaterally
* Measurable transient-evoked otoacoustic emissions
* Ability to read and speak English
* Ability to comply with all test procedures
* Ability to commute to VA Loma Linda Healthcare System 12 times

Exclusion Criteria:

* Hearing asymmetry >15 decibels at three or more audiometric frequencies
* Conductive hearing loss or otologic pathology
* History of middle ear surgery
* Chronic disease and/or use of medication that affects ability to participate in test procedures during study period

Ages: 35 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian B Mertes, PhD, AuD, Principal Investigator — Loma Linda Veterans Association for Research and Education
Locations (1):
- VA Loma Linda Healthcare System, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berlin CI, Hood LJ, Wen H, Szabo P, Cecola RP, Rigby P, Jackson DF. Contralateral suppression of non-linear click-evoked otoacoustic emissions. Hear Res. 1993 Dec;71(1-2):1-11. doi: 10.1016/0378-5955(93)90015-s. PMID 8113128
- [Background] de Boer J, Thornton AR. Neural correlates of perceptual learning in the auditory brainstem: efferent activity predicts and reflects improvement at a speech-in-noise discrimination task. J Neurosci. 2008 May 7;28(19):4929-37. doi: 10.1523/JNEUROSCI.0902-08.2008. PMID 18463246
- [Background] Goodman SS, Mertes IB, Lewis JD, Weissbeck DK. Medial olivocochlear-induced transient-evoked otoacoustic emission amplitude shifts in individual subjects. J Assoc Res Otolaryngol. 2013 Dec;14(6):829-42. doi: 10.1007/s10162-013-0409-9. Epub 2013 Aug 28. PMID 23982894
- [Background] Guinan JJ Jr. Olivocochlear efferents: anatomy, physiology, function, and the measurement of efferent effects in humans. Ear Hear. 2006 Dec;27(6):589-607. doi: 10.1097/01.aud.0000240507.83072.e7. PMID 17086072
- [Background] Mertes IB, Goodman SS. Within- and Across-Subject Variability of Repeated Measurements of Medial Olivocochlear-Induced Changes in Transient-Evoked Otoacoustic Emissions. Ear Hear. 2016 Mar-Apr;37(2):e72-84. doi: 10.1097/AUD.0000000000000244. PMID 26583481
- [Background] Mertes IB, Leek MR. Concurrent measures of contralateral suppression of transient-evoked otoacoustic emissions and of auditory steady-state responses. J Acoust Soc Am. 2016 Sep;140(3):2027. doi: 10.1121/1.4962666. PMID 27914370
- [Background] Miller JD, Watson CS, Kistler DJ, Preminger JE, Wark DJ. Training listeners to identify the sounds of speech: II. Using SPATS software. Hear J. 2008 Oct;61(10):29-33. doi: 10.1097/01.HJ.0000341756.80813.e1. No abstract available. PMID 20209044
- [Result] Mertes IB, Wilbanks EC, Leek MR. Olivocochlear Efferent Activity Is Associated With the Slope of the Psychometric Function of Speech Recognition in Noise. Ear Hear. 2018 May/Jun;39(3):583-593. doi: 10.1097/AUD.0000000000000514. PMID 29135685

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned to Training and Control groups a priori.
Groups:
- Training: Participants in the Training arm will undergo 15 hours of computerized auditory training across 10 laboratory visits. Medial olivocochlear reflex function and speech perception abilities will be measured before, during, and after the training visits to examine the changes in the measurements across time.
  Computerized auditory training: 10 sessions of computerized auditory training (1.5 hr/session) for up to 1 year.
Period: Overall Study
Arm/Group | Training | Control | Speech Group
Started | 10 | 8 | 10
Completed | 5 | 5 | 5
Not Completed | 5 | 3 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Did not meet inclusion criteria | 4 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Training | Control | Speech Group | Total
Number analyzed (Participants) | 10 | 8 | 10 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (5.9) | 63.0 (5.2) | 59.2 (15.4) | 61.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 4
  Male | 10 | 5 | 9 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 9 | 7 | 8 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 0 | 5
  White | 6 | 5 | 8 | 19
  More than one race | 0 | 0 | 2 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 10 | 28
Medial Olivocochlear Reflex Inhibition [Median (Full Range); unit: decibels] — Difference in transient-evoked otoacoustic emission magnitude (in decibels) obtained with versus without presence of contralateral noise. Population: Results are reported for subjects meeting inclusion/exclusion criteria.
  decibels
    number analyzed (Participants) | 5 | 5 | 5 | 15
    (all) | 1.4 [0.8 to 5.1] | 0.6 [-0.01 to 4.0] | 1.9 [1.1 to 4.0] | 1.4 [-0.01 to 5.1]
Performance on Untrained Speech Perception Tasks [Median (Full Range); unit: Percentage correct] — Results obtained on Coordinate Response Measure (CRM) task and Institute of Electrical and Electronics Engineers (IEEE) sentences. CRM and IEEE tasks presented at two decibel signal-to-noise ratios (dB SNR). Results are displayed in percentage correct. Population: Results are displayed for participants meeting inclusion/exclusion criteria.
  Percentage correct
    CRM at -9 dB SNR: number analyzed (Participants) | 5 | 5 | 5 | 15
    CRM at -9 dB SNR | 28 [18 to 42] | 26 [20 to 56] | 28 [8 to 38] | 28 [8 to 56]
    CRM at -6 dB SNR: number analyzed (Participants) | 5 | 5 | 5 | 15
    CRM at -6 dB SNR | 62 [36 to 74] | 58 [52 to 74] | 62 [44 to 66] | 62 [36 to 74]
    IEEE at -6 dB SNR: number analyzed (Participants) | 5 | 5 | 5 | 15
    IEEE at -6 dB SNR | 14 [3 to 36] | 21 [4 to 45] | 17 [12 to 25] | 17 [3 to 45]
    IEEE at -3 dB SNR: number analyzed (Participants) | 5 | 5 | 5 | 15
    IEEE at -3 dB SNR | 62 [14 to 78] | 56 [12 to 80] | 47 [16 to 57] | 56 [12 to 80]

OUTCOME MEASURES:

1. Primary Outcome: Change in Magnitude of Medial Olivocochlear Reflex Inhibition
Description: Decibel difference in medial olivocochlear reflex inhibition computed between final visit and baseline visit, where medial olivocochlear reflex inhibition is quantified as amplitude difference (in decibels) between transient-evoked otoacoustic emissions obtained with versus without broadband noise presented to the contralateral ear.
Time Frame: First and last measurements (baseline and last session up to a year later)
Population: Due to the small sample size in each group, statistical comparisons between groups were not performed. Data were not collected in the Speech Group.
Measure: Median (Full Range); unit: decibel difference
Arm/Group | Training | Control | Speech Group
Number analyzed (Participants) | 5 | 5 | 0
decibel difference | -0.82 [-3.71 to -0.08] | -0.49 [-1.23 to 0.49] |

2. Primary Outcome: Association Between Medial Olivocochlear Reflex Inhibition and Untrained Speech Perception Tasks
Description: Spearman rank correlation computed between medial olivocochlear reflex inhibition (in decibels) and performance (in percent correct) on Coordinate Response Measure (CRM) task and Institute of Electrical and Electronics Engineers (IEEE) sentences, each presented at two decibel signal-to-noise ratios (dB SNR). Results obtained at first study visit.
Time Frame: Baseline (First study visit - 3 hour session)
Population: In order to increase statistical power, the baseline results for medial olivocochlear reflex inhibition results and speech perception from the Training, Control, and Speech Groups were pooled for this analysis
Measure: Number; unit: Spearman Rank Correlation Coefficient
Groups:
- Pooled Participant Data: Baseline data from Training, Control, and Speech Groups pooled together.
Arm/Group | Pooled Participant Data
Number analyzed (Participants) | 15
Spearman Rank Correlation Coefficient
  CRM at -9 dB SNR | -0.18
  CRM at -6 dB SNR | 0.28
  IEEE at -6 dB SNR | -0.06
  IEEE at -3 dB SNR | 0.45
Statistical Analysis 1: Comparison: Pooled Participant Data; Statistical analysis for the row CRM at -9 dB SNR; Test type: Other; p = 0.34, Spearman partial rank correlation; Age and high-frequency pure-tone average controlled for
Statistical Analysis 2: Comparison: Pooled Participant Data; Statistical analysis for the row CRM at -6 dB SNR; Test type: Other; p = 0.64, Spearman partial rank correlation; Age and high-frequency pure-tone average controlled for
Statistical Analysis 3: Comparison: Pooled Participant Data; Statistical analysis for the row IEEE at -6 dB SNR; Test type: Other; p = 0.24, Spearman partial rank correlation; Age and high-frequency average controlled for
Statistical Analysis 4: Comparison: Pooled Participant Data; Statistical analysis for the row IEEE at -3 dB SNR; Test type: Other; p = 0.20, Spearman partial rank correlation; Age and high-frequency average controlled for

3. Secondary Outcome: Change in Auditory Training Sentence Task Performance
Description: Difference in percent correct of auditory training sentences, computed between first and last measurements.
Time Frame: First and last measurements (baseline and last session up to a year later)
Population: Due to the small sample size, statistical analyses of group data were not performed. Data were not collected in the Control or Speech groups.
Measure: Median (Full Range); unit: Difference in percentage correct
Groups:
- Training: Participants in the Training arm will undergo 15 hours of computerized auditory training across 10 laboratory visits. Medial olivocochlear reflex function and speech perception abilities will be measured before, during, and after the training visits to examine the changes in the measurements across time.
  Computerized auditory training: 10 sessions of computerized auditory training (1.5 hr/session) up to 1 year.
Arm/Group | Training
Number analyzed (Participants) | 5
Difference in percentage correct | 3 [-2 to 12]

4. Secondary Outcome: Change in Auditory Training Phoneme Task Performance
Description: Difference in signal-to-noise ratio (in decibels) on auditory training phoneme tasks (onsets, nuclei, and codas), computed between first and last measurement.
Time Frame: First and last measurements (baseline and last session up to a year later)
Population: as for outcome 3
Measure: Median (Full Range); unit: Signal-to-noise ratio change in decibels
Arm/Group | Training
Number analyzed (Participants) | 5
Signal-to-noise ratio change in decibels
  Onsets | -4.38 [-22.98 to -1.99]
  Nuclei | -2.99 [-6.14 to 2.83]
  Codas | -2.60 [-10.99 to 10.37]

5. Post Hoc Outcome: Association Between Medial Olivocochlear Reflex Inhibition and Slope of the Psychometric Function of Untrained Speech Perception Tasks
Description: Partial Spearman rank correlation computed between medial olivocochlear reflex inhibition (in decibels) and slope of the psychometric function (in decibel per decibel) of untrained speech tasks (Coordinate Response Measure -- CRM; Institute of Electrical and Electronics Engineers -- IEEE) obtained from performance across two signal-to-noise ratios. Age and high-frequency pure-tone average were controlled for in this post-hoc analysis. Results obtained at first study visit.
Time Frame: Baseline (First study visit - 3 hour session)
Population: as for outcome 2
Measure: Number; unit: Spearman partial rank correlation
Arm/Group | Pooled Participant Data
Number analyzed (Participants) | 15
Spearman partial rank correlation
  CRM Slope | 0.59
  IEEE Slope | 0.60
Statistical Analysis 1: Comparison: Pooled Participant Data; Statistical analysis for the row CRM slope; Test type: Other; p = 0.03, Spearman partial rank correlation; Age and high-frequency pure-tone average controlled for
Statistical Analysis 2: Comparison: Pooled Participant Data; Statistical analysis for row IEEE slope; Test type: Other; p = 0.04, Spearman partial rank correlation; Age and high-frequency pure-tone average controlled for

ADVERSE EVENTS:
Time Frame: Through study completion, maximum of 1 year.
Description: Definition of adverse event and/or serious adverse event are consistent with clincialtrials.gov definitions.
Arm/Group | Training | Control | Speech Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/8 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Training (N=10) | Control (N=8) | Speech Group (N=10)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT02574247/Prot_SAP_001.pdf